CLINICAL TRIAL: NCT05340777
Title: GHANA: An Implementation Study on the Barriers and Facilitators of Scaling up the Innovative, Low-cost Ellavi Uterine Balloon Tamponade for Postpartum Hemorrhage
Brief Title: Ghana: The Barriers and Facilitators of Scaling up the Ellavi UBT for Postpartum Hemorrhage
Status: Completed | Type: Observational
Sponsor: PATH (Other)
Collaborators: Ghana Health Services (Other Government)
Responsible Party: Principal Investigator, Megan Parker, Senior Research Officer, PATH
Other Study IDs: 1514537
Record Dates: First submitted 2021-09-14; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Training Obstetric staff on Ellavi UBT — The study team will train all obstetric healthcare staff (i.e. obstetricians, midwives, medical officers, clinical officers) involved in PPH management at the participating healthcare facilities on use of the Ellavi UBT. This will be done to ensure staff are trained on the newly registered and provided medical device. We will gather feedback on how to improve the training curriculum from participants. We will also gather information from the healthcare workers immediately post-use of an Ellavi UBT device following their management of a refractory PPH case. These surveys will help us to understand the barriers to and facilitators of use in order to evaluate acceptability and feasibility among facilities providing different levels of PPH care.

SUMMARY:
The purpose of this implementation science study is to generate evidence that informs the successful uptake and adoption of the Ellavi UBT within Ghana's PPH management programs. The investigators aim to improve the likelihood that the Ellavi UBT will be integrated into the health care system by obtaining critical feedback from stakeholders and health care providers on the barriers and facilitators towards its successful adoption and roll out. The research will be done in three purposively selected facilities near Accra Ghana: Tema General Hospital, Ridge Hospital, and Kasoa Polyclinic.

This study uses a nonexperimental design to collect data on implementation (e.g. # staff trained, usability, user confidence, acceptability, feasibility). The study team will train all obstetric healthcare staff (i.e. obstetricians, midwives, medical officers, clinical officers) involved in PPH management at the 3 participating healthcare facilities on the Ellavi UBT. The investigators will gather feedback from the obstetric healthcare workers (post-training and post-PPH) to understand the barriers to and facilitators of use in order to evaluate acceptability and feasibility among facilities providing different levels of care (level 4, level 5 (county), level 6 (tertiary)). This process will help to generate training and facility level recommendations for improved uptake and integration into the local maternal care package. Case report forms and semi-quantitative surveys will be completed by obstetrical care providers to evaluate the primary outcomes of acceptability and feasibility by measuring: context of use, accuracy of use, perceptions of the device, user confidence, acceptability, usability, facilitators of use, barriers to use, use-patterns, and insights into training effectiveness. The secondary outcomes will include financial data to determine the cost of introducing the Ellavi UBT into the Kenyan PPH management protocols and the health system. The study will not involve the storage of biological samples. There is not a direct benefit of the study to the individual participants. All study participants will sign consent forms.

DETAILED DESCRIPTION:
The purpose of this implementation research study is to generate evidence that informs the successful uptake and adoption of the Ellavi UBT within Ghanaian PPH management programs for both public and private sector programs. The investigators aim to generate evidence for Ghanaian stakeholders to use in their decision-making around the use of Ellavi UBT in PPH management programs.

Specific objectives:

To determine the adoption, penetration, sustainability and fidelity of implementing the Ellavi UBT device into PPH care in three health care facilities. The investigators will explore the number of health workers and facilities that receive the PPH and Ellavi UBT training, and percent of health workers and facilities that adopt the Ellavi UBT device over the 10-month period. The investigators will also assess factors that influence the adoption, penetration, sustainability, and fidelity through an operations research survey, and the Ellavi UBT questionnaire.

To determine the appropriateness, acceptability and feasibility of using the Ellavi UBT in participating health facilities at various levels of care near Accra, the investigators will explore user comprehension of the Ellavi UBT usage steps, accuracy of use, perceptions of the device, attitudes towards the device, user confidence, usability, facilitators of use, barriers to use, use-patterns, and insights into training effectiveness.

* Sensitize senior management at each of the three participating facilities, separately.
* Conduct two half-day trainings on PPH and Ellavi UBT use at each of the three participating health facilities separated by: 1) obstetricians, medical and clinical officers, and 2) midwives.
* Collect individual initial (post-training) data to assess comprehension of Ellavi UBT usage steps, perceptions of the device, attitudes towards the device, user confidence, usability, and insights into training effectiveness.
* Case Management Form (CMF): Obstetrical care provider will complete a CMF within 24hrs (<24hrs) of managing each PPH event. This will inform the study team of how decision-making algorithms were applied and accuracy of use.
* Ellavi UBT Questionnaire: PATH-Ghana study team member will collect individual post (post-usage) Ellavi UBT use data (<72hrs) from each study participant (obstetrical care worker) to assess comprehension of Ellavi UBT usage steps, perceptions of the device, attitudes towards the device, user confidence, usability, facilitators of use, barriers to use, use-patterns, and insights into training effectiveness.
* PATH-Ghana study staff will record secondary data from hospital registry books over a 9 month duration of this study (January-Sept 2021) in comparison to the same period in 2020 to examine changes in use of condom catheters, and Ellavi UBTs.
* Use the Consolidated Framework for Implementation Research (CFIR) to identify constructs with the potential to influence the introduction and use of Ellavi UBT. These constructs will be mapped to questions in the questionnaire, and will be analyzed to identify their influence on Ellavi UBT use. Constructs that have influence on the implementation of UBTs (both positively and negatively) will be disseminated for use in future introduction and scale up of Ellavi UBTs.

To disseminate the information in national, regional, and international forums to support information sharing, increased awareness of the role of UBT for refractory PPH, and adoption of its use.

* Summarize how the Ellavi UBT can be integrated into curriculums, guidelines, and hospital systems (e.g. patient-provider friendly materials) by analyzing the key facilitators and barriers.
* Host a national level meeting with Kenyan MOH stakeholders and participating facilities
* Publish and disseminate findings in a peer-reviewed journal h. Present at international conferences and forums, as funding permits. Show the use of Ellavi UBT using poster presentations and demonstration sessions at international obstetrics meetings: FIGO, WHO UBT group, Women Deliver as funding permits.

ELIGIBILITY:
Inclusion Criteria:

* Labor ward obstetric staff
* Employed at 1 of the 3 hospitals participating in this study.

Exclusion Criteria:

* Non-obstetric staff
* Obstetric staff not employed at the 3 study hospitals

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Obstetrical care providers who recently participated in a PPH/Ellavi UBT training and/or obstetrical care providers who recently managed a refractory PPH event. The study participant must work in 1 of 3 participating facilities. The number of interviewees per site will vary depending on the size of the facility and number of refractory PPH events.
  Participants will be selected based on their participation in training sessions, or their management of a PPH event and will include obstetrical staff currently practicing at Tema General Hospital, Kasoa Polyclinic, or Ridge Hospital. Participants may be re-sampled with each use of the UBT.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Semi-quantitative post-training survey on the appropriateness and acceptability of using the Ellavi UBT device | 10 months
  * Appropriateness will be measured by capturing # deliveries and # postpartum hemorrhage (PPH) cases typically managed per month by the obstetric staff surveyed.
  * Acceptability will be measured by surveying obstetric staff on their perception of Ellavi UBT effectiveness in comparison to other PPH treatments, attitudes towards the device post training, device usability measures, and user-confidence operating the device.
Facility survey (quantitative) to determine adoption, penetration, and sustainability | 10 months
  * Adoption will be measured by the # of facilities (of 3 total) who ever used the Ellavi UBT over the 10 month period.
  * Penetration/Reach will be measured by determining the % of total staff (employed at the 3 hospitals) who were participated in our Ellavi UBT/PPH training courses.
  * Sustainability is measured by the # facilities (of 3 total) who ever used the Ellavi UBT 4 months after the training (at least 1 time), and the # of facilities that used the Ellavi UBT every month for 6 months after the training.
Semi-quantitative post-UBT-use survey on fidelity to training skills, and feasibility of using the Ellavi UBT device | 10 months
  * Feasibility will be measured by capturing the # of Ellavi UBT devices used to manage the PPH events, and barriers/enablers to use of the device.
  * Fidelity will be measured by questions asked on accuracy of use (fidelity to the training)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Parker, PhD, Principal Investigator — PATH
Locations (3):
- Ghana (3):
  - Kasoa Polyclinic, Kasoa, Central Region
  - Ridge Hospital, Accra
  - Tema General Hospital, Accra

IPD SHARING:
Plan to Share IPD: No
The de-identified data will be shared with the funder in the form of a study report. If data are held on a public database (due to publication requirements), they will not be linked to the study participant and their identity would not be revealed.

REFERENCES:
- [Derived] Parker ME, Qureshi Z, Deganus S, Soki J, Cofie P, Dapaah P, Owusu R, Gwako G, Osoti A, Ogutu O, Opira J, Sunkwa-Mills G, Boamah M, Srofenyoh E, Aboagye P, Fofie C, Kaliti S, Morozoff C, Secor A, Metzler M, Abu-Haydar E. Introduction of the Ellavi uterine balloon tamponade into the Kenyan and Ghanaian maternal healthcare package for improved postpartum haemorrhage management: an implementation research study. BMJ Open. 2023 Feb 3;13(2):e066907. doi: 10.1136/bmjopen-2022-066907. PMID 36737079